CLINICAL TRIAL: NCT03400228
Title: Effect of Probiotic Consumption on Chronic Kidney Disease and Cardiovascular Risk
Brief Title: Effect of Probiotic Consumption on Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Univates (Other)
Responsible Party: Principal Investigator, Thaís Rodrigues Moreira, Principal Investigator, Centro Universitário Univates
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 072015
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Chronic Kidney Disease
Keywords: Probiotics; Chronic kidney disease; Cardiovascular risk
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protics (Experimental): Patients in the intervention group were to drink 2 sachets of 1g of probiotic daily for 24 weeks
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Patients in the intervention group were to drink 2 sachets of 1g of maltodextrin daily for 24 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotic — The probiotic is composed of a combination of Lactobacillus acidophilus (LA-5®) and Bifidobacterium lactis (BB-12®).
  Arms: Protics
Dietary Supplement: Maltodextrin — Maltodextrin is a supplement feed based carbohydrate powder and tasteless.
  Arms: Placebo

SUMMARY:
Recent studies have demonstrated that the balance of intestinal microbiota is affected in chronic kidney disease (CKD), leading to a condition known as intestinal dysbiosis. These changes were associated with metabolic complications, accumulation of uremic toxins, inflammation, progression of CKD and cardiovascular risk. Measures with the aim of restore the balance of intestinal flora are suggested, such as the intake of probiotics composed of beneficial bacteria, but few studies have discussed the effect of these supplements in CKD. The present study aims to evaluate the effect of consumption of probiotics in factors associates with progression of CKD and cardiovascular risk. To such will be conducted a double-blind, placebo-controlled, and randomized clinical trial with 30 patients with CKD in stages 3-5, treated in ambulatories of Nephrology of the Hospital de Clínicas de Porto Alegre, independently of etiology and with steady renal function. Patients will be excluded whether in substitutive renal therapy, kidney transplant, on antimicrobial therapy or immunosuppressive agents in the last three months or with acute clinical events. The assessment will include clinical and nutritional parameters, estimated glomerular filtration rate, proteinuria, serum lipids, inflammatory factors, and bowel habits. The study protocol includes the recruitment of patients who will undergo to 4-week washout period. After patients will be randomized and provided with probiotic therapy (intervention group) or placebo (maltodextrin; control group) for 24 weeks. All patients will be instructed to consume 2 sachets/day of probiotic or placebo and receive nutritional advice. All data will be analysed by the principal investigator with the support of a trained statistician and the chief investigator. The statistical programme SPSS will be used.

DETAILED DESCRIPTION:
The assessment will include clinical and nutritional parameters, estimated glomerular filtration rate, proteinuria, serum lipids, inflammatory factors, and bowel habits. The study protocol includes the recruitment of patients who will undergo to 4-week washout period. After patients will be randomized and provided with probiotic therapy (intervention group) or placebo (maltodextrin; control group) for 24 weeks. All patients will be instructed to consume 2 sachets/day of probiotic or placebo and receive nutritional advice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease stage 3, 4 and 5;
* Stable renal function;
* Proteinuria greater than or equal to 500 mg;
* Patients who agree to participate.

Exclusion Criteria:

* Patients on renal replacement therapy or kidney transplant;
* Patients with prior renal transplant;
* Patients with acute clinical events;
* Patients using antibiotics or any other medications that can alter the intestinal microbiota as corticosteroids and immunosuppressants in the last three months;
* Patients with active infection;
* Patients with inflammatory bowel diseases or malabsorption;
* Acute or chronic diarrhea;
* Patients with previous intestinal surgery;
* Pregnants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Decrease in serum creatinine level | 24 weeks
  Reduction of serum creatinine level

SECONDARY OUTCOMES:
Reduced levels of serum lipids | 24 weeks
  Reduced serum cholesterol level

CONTACTS AND LOCATIONS:
Overall Officials: Thais Rodrigues, Moreira, Principal Investigator — university
Locations (1):
- Thaís Rodrigues Moreira, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
There is no plan to make available individual participant data (IPD) to other researchers.